CLINICAL TRIAL: NCT06172309
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetics and Preliminary Pharmacodynamic Effect of NTQ1062 Tablets in Chinese Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of NTQ1062 in Chinese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTQ1062-21101
Record Dates: First submitted 2023-11-23; First posted 2023-12-15 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NTQ1062 (Experimental): NTQ1062 Tablets will be administered orally QD in a 28-day cycle (21 days on treatment followed by 7 days off treatment) in sequential cohorts.
  Interventions: Drug: NTQ1062

INTERVENTIONS:
Drug: NTQ1062 — tablet(s) PO

SUMMARY:
This is an open-label, single-arm, phase 1 study to evaluate the safety, tolerability, pharmacokinetics, and preliminary pharmacodynamic effect of NTQ1062 in patients with advanced solid tumors.

The study comprises a dose-escalation phase and a dose-expansion phase.

1. Dose-escalation:using 3+3 design to evaluate the safety, tolerability, and pharmacokinetic profile of NTQ1062 at 20, 50, 100, 200, 300, 400 mg in patients with advanced solid tumors, and to determine the maximum tolerated dose (MTD).
2. Dose-expansion:the dose-expansion study will evaluate the safety, tolerability, and preliminary pharmacodynamic effect of the MTD for NTQ1062 in patients with advanced solid tumors, and to identify the recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years old, male or female patients.
2. Patients with histologically and cytologically confirmed, advanced malignant solid tumors who have progressed on standard therapy or for whom no standard therapy exists, or for whom no standard treatment is available.
3. (Dose escalation phase)Solid tumors that are at least one evaluable per Response Evaluation Criteria in Solid Tumors(RECIST v1.1);(Dose expansion phase)Solid tumors that are at least one measurable per Response Evaluation Criteria in Solid Tumors(RECIST v1.1).
4. ECOG score is 0-1.
5. Predicted life expectancy ≥3 months.
6. Patients must have adequate organ function:

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet count ≥ 75×109/L, hemoglobin ≥ 85 g/L.
   2. Liver function: Total bilirubin ≤ 1.5xULN, AST and ALT ≤ 3.0xULN (≤ 5.0xULN for patients with Patients with hepatic metastases or hepatic carcinoma).
   3. Renal function:Creatinine (Cr) ≤ 1.5xULN or creatinine clearance (Ccr) ≥ 50 ml/min/1.73m2.
   4. Coagulation function: activated partial thromboplastin time (APTT) and INR ≤1.5×ULN.
7. Female patients of child-bearing potential, and all male partners must consent to use a acceptable method of contraception throughout the study period and for 90 days after the last dose of either study drug.
8. Patients must be signed written informed consent prior to admission to the study.

Exclusion Criteria:

1. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   1. Diagnosis of diabetes mellitus type I.
   2. Baseline fasting glucose value of ≥8.33 mmol/l (150 mg/dL).
   3. Glycosylated haemoglobin (HbA1C) ≥8%.
2. Patients who are still receive anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor drug from 4 weeks prior to the first dose.
3. Patients have received previous treatment with a AKT,PI3K or mTOR inhibitor.
4. Patients received strong inhibitors and/or inducers of CYP3A4 within 7 days prior to the first dose of study drug.
5. Active infection requiring systemic treatment.
6. Active hepatitis B virus infection or hepatitis C virus infection.
7. History of human immunodeficiency virus infection.
8. Patient has symptomatic CNS metastases.
9. History of severe cardiovascular diseases.
10. Other conditions that the investigator considers inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | First treatment cycle (i.e., the first 28 days post the first dose)
  The MTD is defined as the highest dose reached for which the incidence of dose limiting toxicity (DLT) occurs in less than 1/3 of the subjects.
Recommended phase 2 dose (RP2D) | First treatment cycle (i.e., the first 28 days post the first dose)
  The RP2D of NTQ1062 will be determined during the dose-escalation phase of the study. RP2D will be determined using available safety and pharmacokinetics and pharmacodynamics data.
Adverse events | through study completion, an average of 1 year
  Safety and tolerability of NTQ1062. Incidence of adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic parameters:Cmax | At the end of Cycle 1 (each cycle is 28 days)
  Maximum Serum Concentration (Cmax) of NTQ1062.
Pharmacokinetic parameters: Tmax | At the end of Cycle 1 (each cycle is 28 days)
  Time to Maximum Serum Concentration (Tmax) of NTQ1062.
Pharmacokinetic parameters: AUC | At the end of Cycle 1 (each cycle is 28 days)
  The area under the concentration versus time curve of NTQ1062.
Pharmacokinetic parameters:T1/2 | At the end of Cycle 1 (each cycle is 28 days)
  The terminal half-life of NTQ1062.
Objective response rate (ORR) | through study completion, an average of 1 year
  ORR is defined as participants with confirmed complete or partial response (CR+PR) per RECIST, v1.1
Disease Control Rate(DCR) | through study completion, an average of 1 year
  DCR was defined as the proportion of patients who had an overall response of complete response (CR), partial response (PR), or stable disease (SD).
Duration of Response(DOR) | through study completion, an average of 1 year
  DOR is defined as the time between date of first response and the first occurrence. of progression or death from any cause, whichever occurs first.
Progression-free Survival(PFS) | through study completion, an average of 1 year
  PFS will be defined as the time between the first dose of any study drug and the first occurrence of progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No